CLINICAL TRIAL: NCT05247229
Title: Prevention of Paralytic Shellfish Poisoning in Subsistence Shellfish Harvest Communities of Southeast Alaska
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Matthew O'Madigan Gribble, Principal Investigator, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 300006786; R01ES029165 (NIH)
Record Dates: First submitted 2022-01-31; First posted 2022-02-18 (Actual); Results first posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Shellfish Poisoning, Paralytic
MeSH Terms: conditions — Shellfish Poisoning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Middle school education program (Experimental): The education intervention centered around teaching children about local traditional ecological knowledge and traditional harvesting and gathering practices, including those for shellfish.
  The education program was divided into three units, following other tribal education programs. Primary data collection was conducted by unit to assess student learning for each unit. The first unit covered an introduction to shellfish, harmful algal blooms (HAB), and paralytic shellfish poisoning (PSP). The second unit covered herring, and how herring relates to Tlingit culture. The third unit focused on intertidal zones as they relate to Tlingit culture.
  Interventions: Behavioral: Middle school education program

INTERVENTIONS:
Behavioral: Middle school education program — The intervention assessed the impact of a middle school education program (implemented as an after school program in Sitka, AK and Juneau, AK and during school hours as an elective in Hoonah, AK) on shellfish and toxin knowledge and clam harvesting planned behaviors. The intervention took place weekly during the school year. The curriculum centered around teaching children about local traditional ecological knowledge and traditional harvesting and gathering practices.

SUMMARY:
The purpose of this tribally co-led community-based participatory research in partnership with Sitka Tribe of Alaska was to help prevent Paralytic Shellfish Poisoning (PSP) in children of Southeast Alaska. The investigators assessed whether an education intervention led to changes in participants' planned behaviors related to clam harvesting that may reduce risks of exposure to shellfish toxins. This project included both a human subjects research component (this clinical trial) and a non-human environmental research component. In the non-human component, the tribe monitored for toxins in shellfish (including shellfish provided by people with data originally collected as a non-research service), and tested water for the presence of algae that make the toxin. The human subjects component involved age-appropriate K12 educational outreach in partnership with the Sitka School District, Hoonah City Schools, and Juneau School District, including a middle school after-school non-credit educational program coupled to a research program in Sitka, AK and Juneau, AK; and a middle school during school elective educational program coupled to a research program in Hoonah, AK. Middle school students participating in the program attended the program with several units designed to teach cultural practices, strengthen competencies toward Alaska science state standards, and evaluate shellfish consumption-related risk behaviors, while affirming traditional culture.

DETAILED DESCRIPTION:
Subsistence use of natural resources, including the subsistence harvesting of shellfish, is central to Native cultures throughout Alaska. Shellfish harvesting appears as a motif in form line artwork and is a part of the traditional food ways taught by the tribes of Southeast Alaska to their youth. Saxitoxin, a toxin detected in Southeast Alaska that causes paralytic shellfish poisoning (PSP), was named after the butter clam (Saxidomus gigantea), which is a traditional food staple. The culturally central consumption of non-commercial shellfish puts Alaska Native communities at elevated risk for PSP. A population-based survey in two communities in coastal Alaska found that 20% of Alaska Natives in their sample reported a history of PSP.

The Theory of Planned Behavior is a behavioral science framework that has been applied in numerous public health settings to understand why people pursue specific actions. The Theory of Planned Behavior has been applied to children's health and to poisoning prevention/ environmental health, but as far as the investigators are aware this is the first pediatric poisoning prevention application of this framework. The project's K12 programming was developed with this framework in mind. For the middle school research program (this clinical trial), the investigators aimed to measure the relevant constructs for a theory-based investigation into children's poisoning-related risk behaviors in a context that affirms safe practice of cultural traditions.

ELIGIBILITY:
Inclusion Criteria:

* Middle school student at Blatchley Middle School in Sitka, Alaska or middle school student at Hoonah City Schools in Hoonah, Alaska or middle school student at Dzantik'i Heeni Middle School in Juneau, Alaska

Exclusion Criteria:

* Not middle school student at Blatchley Middle School in Sitka, Alaska or middle school student at Hoonah City Schools in Hoonah, Alaska or middle school student at Dzantik'i Heeni Middle School in Juneau, Alaska

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Hoonah City Schools, Hoonah, Alaska
  - Dzantik'i Heeni Middle School, Juneau, Alaska
  - Sitka Tribe of Alaska, Sitka, Alaska

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roland HB, Kohlhoff J, Moore TR, Lanphier K, Pierce L, Narvaez J, Yazzie A, Whitehead C, Feldpausch J, Gribble MO. Influence of a Tribally Led Children's Environmental Education Program on Shellfish Harvesting Beliefs and Behavioral Intentions. Community Sci. 2025 Sep;4(3):e2025CSJ000128. doi: 10.1029/2025CSJ000128. Epub 2025 Sep 3. PMID 41574333

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants who enrolled in the study completed the study.
Groups:
- Middle School Education Program: The education intervention centers around teaching children about local traditional ecological knowledge and traditional harvesting and gathering practices, including those for shellfish.
  The education program is divided into three units, following other tribal education programs. Primary data collection will be conducted by unit to assess student learning for each unit. The first unit will cover an introduction to shellfish, harmful algal blooms (HAB), and paralytic shellfish poisoning (PSP). The second unit will cover herring and how herring relates to Tlingit culture. The third unit will focus on intertidal zones as zones relate to Tlingit culture.
Period: Overall Study
Arm/Group | Middle School Education Program
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The overall number of baseline participants is the same as the number assigned to the single arm.
Arm/Group | Middle School Education Program
Number analyzed (Participants) | 50
Age, Continuous [Mean (Full Range); unit: years] | 12.6 [11 to 14]
Sex/Gender, Customized [Count of Participants; unit: Participants] — Sex/ Gender: Male, Female, Nonbinary, Questioning, Not reported (response options included an open ended option; not all participants reported their sex/ gender).
  Participants
    Male | 21
    Female | 18
    Nonbinary | 5
    Questioning | 1
    Not reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 9
  More than one race | 25
  Unknown or Not Reported | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 3
Pre-program survey responses [Mean (Standard Deviation); unit: Scores on a scale] — Likert-scale responses ranging from disagree (1) to agree (5) Population: Differences between the participant numbers in the rows and the overall numbers are due to participant non-response.
  Scores on a scale
    1: Subsistence clam harvesting is enjoyable: number analyzed (Participants) | 39
    1: Subsistence clam harvesting is enjoyable | 3.6 (0.9)
    2: Subsistence clam harvesting is rewarding: number analyzed (Participants) | 39
    2: Subsistence clam harvesting is rewarding | 4.1 (1.0)
    3: People I care about approve of clam harvest: number analyzed (Participants) | 43
    3: People I care about approve of clam harvest | 4.3 (1.0)
    4: Peers participate in clam harvesting: number analyzed (Participants) | 43
    4: Peers participate in clam harvesting | 3.1 (1.2)
    5: Whether I harvest is up to me: number analyzed (Participants) | 43
    5: Whether I harvest is up to me | 4.2 (1.2)
    6: I intend to clam harvest this year: number analyzed (Participants) | 43
    6: I intend to clam harvest this year | 4.0 (1.3)
    7: I have participated in clam harvesting: number analyzed (Participants) | 42
    7: I have participated in clam harvesting | 2.5 (1.8)
    9: Checking website before clamming is rewarding: number analyzed (Participants) | 37
    9: Checking website before clamming is rewarding | 3.5 (1.3)
    10: Checking website before clamming is easy: number analyzed (Participants) | 37
    10: Checking website before clamming is easy | 3.8 (1.2)
    11: Those I get clams with approve of check site: number analyzed (Participants) | 35
    11: Those I get clams with approve of check site | 3.9 (1.2)
    12: People like me will check website before clam: number analyzed (Participants) | 37
    12: People like me will check website before clam | 3.2 (1.3)
    13: I am confident I can check website before clam: number analyzed (Participants) | 38
    13: I am confident I can check website before clam | 3.6 (1.2)
    14: Checking website is up to me: number analyzed (Participants) | 38
    14: Checking website is up to me | 4.0 (1.2)
    15: I intend to check website to decide to clam: number analyzed (Participants) | 38
    15: I intend to check website to decide to clam | 3.8 (1.2)
Pre-program interview themes [Count of Participants; unit: Participants] — Population: Differences between the participant numbers in the rows and the overall numbers are due to 37 total pre-program interviews being conducted with participants.
  Participants
    Some/ high knowledge of PSP: number analyzed (Participants) | 37
    Some/ high knowledge of PSP | 15
    Some/ high knowledge of risk reduction strategies: number analyzed (Participants) | 37
    Some/ high knowledge of risk reduction strategies | 8
    Some/ high knowledge of SEATOR resources: number analyzed (Participants) | 37
    Some/ high knowledge of SEATOR resources | 3

OUTCOME MEASURES:

1. Primary Outcome: Student Assessment Questionnaire of Student Learning From Each Educational Unit.
Description: The investigators will assess student learning with pre-unit and post-unit written evaluations that collect information on students' cultural and scientific knowledge using Likert scale questions. Likert-scale responses ranged from disagree (1) to agree (5). Here we report post education unit outcomes. We report pre education unit outcomes in baseline characteristics. Questions 10 and 13 of our survey reflect this outcome measure.
Time Frame: The time frame is one educational semester, lasting 10 weeks (10 units administered weekly). Here we report post education unit outcomes (following the semester-long program). We report pre education program outcomes in baseline characteristics.
Population: Differences between the population numbers in the rows and the overall numbers are due to participant non-response.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Middle School Education Program
Number analyzed (Participants) | 50
Scores on a scale
  10: Checking website before clamming is easy: number analyzed (Participants) | 48
  10: Checking website before clamming is easy | 4.2 (0.9)
  13: I am confident I can check website before clam: number analyzed (Participants) | 48
  13: I am confident I can check website before clam | 3.9 (1.3)
Statistical Analysis 1: Comparison: Middle School Education Program; Q10 Difference between pre- and post-program surveys from generalized estimating equation linear regressions accounting for clustering of longitudinal observations within person, adjusted associations and 95% confidence intervals; Test type: Superiority; p = 0.05, Chi-squared; Slope = 0.37, 95% CI 2-sided [0.00 to 0.73]
Statistical Analysis 2: Comparison: Middle School Education Program; Q13 Difference between pre- and post-program surveys from generalized estimating equation linear regressions accounting for clustering of longitudinal observations within person, adjusted associations and 95% confidence intervals; Test type: Superiority; p = 0.36, Chi-squared; Slope = 0.22, 95% CI 2-sided [-0.25 to 0.70]

2. Primary Outcome: Student Assessment Questionnaire of Student Behaviors and Behavioral Intentions Related to Shellfish Consumption and Checking SEATOR Website (Accessing a Tribal Resource to Prevent Poisoning).
Description: The investigators will assess changes in student self-reported behavioral history and student behavioral intentions with pre-unit and post-unit written evaluations that collect information on students' history to date of participating in subsistence shellfish harvest activities and students' behavioral intentions to participate in subsistence shellfish harvest activities and to check the SEATOR website, measured using Likert scale questions. Likert-scale responses ranged from disagree (1) to agree (5). Here we report post education unit outcomes. We report pre education unit outcomes in baseline characteristics. Questions 6, 7, 8, 15, and 16 reflect this outcome measure. Questions 8 and 16 are excluded from the pre-post program statistical tests as these questions are only relevant in the post-program survey.
Time Frame: as for outcome 1
Population: Differences between the population numbers in the rows and the overall numbers are due to participant non-response.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Middle School Education Program
Number analyzed (Participants) | 50
Scores on a scale
  6: I intend to clam harvest this year: number analyzed (Participants) | 47
  6: I intend to clam harvest this year | 3.4 (1.4)
  7: I have participated in clam harvesting: number analyzed (Participants) | 47
  7: I have participated in clam harvesting | 2.8 (1.8)
  8: Learning clam safety I am more willing to clam: number analyzed (Participants) | 47
  8: Learning clam safety I am more willing to clam | 4.4 (0.9)
  15: I intend to check website to decide to clam: number analyzed (Participants) | 47
  15: I intend to check website to decide to clam | 3.9 (1.0)
  16: I have used website to inform decision to clam: number analyzed (Participants) | 47
  16: I have used website to inform decision to clam | 3.1 (1.5)
Statistical Analysis 1: Comparison: Middle School Education Program; Q6 Difference between pre- and post-program surveys from generalized estimating equation linear regressions accounting for clustering of longitudinal observations within person, adjusted associations and 95% confidence intervals; Test type: Superiority; p = 0.12, Chi-squared; Slope = -0.42, 95% CI 2-sided [-0.96 to 0.11]
Statistical Analysis 2: Comparison: Middle School Education Program; Q7 Difference between pre- and post-program surveys from generalized estimating equation linear regressions accounting for clustering of longitudinal observations within person, adjusted associations and 95% confidence intervals; Test type: Superiority; p = 0.21, Chi-squared; Slope = 0.41, 95% CI 2-sided [-0.23 to 1.05]
Statistical Analysis 3: Comparison: Middle School Education Program; Q15 Difference between pre- and post-program surveys from generalized estimating equation linear regressions accounting for clustering of longitudinal observations within person, adjusted associations and 95% confidence intervals; Test type: Superiority; p = 0.78, Chi-squared; Slope = 0.07, 95% CI 2-sided [-0.41 to 0.54]

3. Primary Outcome: Student Assessment Questionnaire of Feelings About Shellfish Harvesting Relevant to the Theory of Planned Behavior.
Description: The investigators will assess changes in student self-reported feelings about shellfish harvesting relevant to the Theory of Planned Behavior, including whether students think shellfish harvesting is enjoyable and rewarding, whether peers approve of shellfish harvesting and participate in shellfish harvesting, and whether students feel empowered to make shellfish harvesting decisions, with pre-unit and post-unit written evaluations that collect information on students' feelings about shellfish harvesting, measured using Likert scale questions. Likert-scale responses ranged from disagree (1) to agree (5). Here we report post education unit outcomes. We report pre education unit outcomes in baseline characteristics. Questions 1, 2, 3, 4, 5, 9, 10, 11, 12, 13, and 14 reflect this outcome measure. Questions 10 and 13 are used to assess both this outcome and primary outcome 1 and so are reported under both measures.
Time Frame: as for outcome 1
Population: Differences between the population numbers in the rows and the overall numbers are due to participant non-response.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Middle School Education Program
Number analyzed (Participants) | 50
Scores on a scale
  1: Subsistence clam harvesting is enjoyable: number analyzed (Participants) | 48
  1: Subsistence clam harvesting is enjoyable | 4.2 (0.8)
  2: Subsistence clam harvesting is rewarding: number analyzed (Participants) | 47
  2: Subsistence clam harvesting is rewarding | 4.2 (1.0)
  3: People I care about approve of clam harvest: number analyzed (Participants) | 48
  3: People I care about approve of clam harvest | 4.4 (0.7)
  4: Peers participate in clam harvesting: number analyzed (Participants) | 48
  4: Peers participate in clam harvesting | 3.1 (1.2)
  5: Whether I harvest is up to me: number analyzed (Participants) | 47
  5: Whether I harvest is up to me | 4.4 (0.7)
  9: Checking website before clamming is rewarding: number analyzed (Participants) | 48
  9: Checking website before clamming is rewarding | 4.3 (0.8)
  10: Checking website before clamming is easy: number analyzed (Participants) | 48
  10: Checking website before clamming is easy | 4.2 (0.9)
  11: Those I get clams with approve of check site: number analyzed (Participants) | 48
  11: Those I get clams with approve of check site | 4.3 (0.9)
  12: People like me will check website before clam: number analyzed (Participants) | 48
  12: People like me will check website before clam | 3.5 (1.3)
  13: I am confident I can check website before clam: number analyzed (Participants) | 48
  13: I am confident I can check website before clam | 3.9 (1.3)
  14: Checking website is up to me: number analyzed (Participants) | 48
  14: Checking website is up to me | 4.4 (1.0)
Statistical Analysis 1: Comparison: Middle School Education Program; Q1 Difference between pre- and post-program surveys from generalized estimating equation linear regressions accounting for clustering of longitudinal observations within person, adjusted associations and 95% confidence intervals; Test type: Superiority; p = 0.01, Chi-squared; Slope = 0.51, 95% CI 2-sided [0.16 to 0.86]
Statistical Analysis 2: Comparison: Middle School Education Program; Q2 Difference between pre- and post-program surveys from generalized estimating equation linear regressions accounting for clustering of longitudinal observations within person, adjusted associations and 95% confidence intervals; Test type: Superiority; p = 0.67, Chi-squared; Slope = 0.09, 95% CI 2-sided [-0.34 to 0.52]
Statistical Analysis 3: Comparison: Middle School Education Program; Q3 Difference between pre- and post-program surveys from generalized estimating equation linear regressions accounting for clustering of longitudinal observations within person, adjusted associations and 95% confidence intervals; Test type: Superiority; p = 0.35, Chi-squared; Slope = 0.13, 95% CI 2-sided [-0.15 to 0.41]
Statistical Analysis 4: Comparison: Middle School Education Program; Q4 Difference between pre- and post-program surveys from generalized estimating equation linear regressions accounting for clustering of longitudinal observations within person, adjusted associations and 95% confidence intervals; Test type: Superiority; p = 0.73, Chi-squared; Slope = 0.09, 95% CI 2-sided [-0.43 to 0.61]
Statistical Analysis 5: Comparison: Middle School Education Program; Q5 Difference between pre- and post-program surveys from generalized estimating equation linear regressions accounting for clustering of longitudinal observations within person, adjusted associations and 95% confidence intervals; Test type: Superiority; p = 0.23, Chi-squared; Slope = 0.20, 95% CI 2-sided [-0.13 to 0.52]
Statistical Analysis 6: Comparison: Middle School Education Program; Q9 Difference between pre- and post-program surveys from generalized estimating equation linear regressions accounting for clustering of longitudinal observations within person, adjusted associations and 95% confidence intervals; Test type: Superiority; p = 0.00, Chi-squared; Slope = 0.71, 95% CI 2-sided [0.27 to 1.15]
Statistical Analysis 7: Comparison: Middle School Education Program; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.05, Chi-squared; Slope = 0.37, 95% CI 2-sided [0.00 to 0.73]
Statistical Analysis 8: Comparison: Middle School Education Program; Q11 Difference between pre- and post-program surveys from generalized estimating equation linear regressions accounting for clustering of longitudinal observations within person, adjusted associations and 95% confidence intervals; Test type: Superiority; p = 0.10, Chi-squared; Slope = 0.37, 95% CI 2-sided [-0.07 to 0.82]
Statistical Analysis 9: Comparison: Middle School Education Program; Q12 Difference between pre- and post-program surveys from generalized estimating equation linear regressions accounting for clustering of longitudinal observations within person, adjusted associations and 95% confidence intervals; Test type: Superiority; p = 0.32, Chi-squared; Slope = 0.30, 95% CI 2-sided [-0.30 to 0.91]
Statistical Analysis 10: Comparison: Middle School Education Program; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.36, Chi-squared; Slope = 0.22, 95% CI 2-sided [-0.25 to 0.70]
Statistical Analysis 11: Comparison: Middle School Education Program; Q14 Difference between pre- and post-program surveys from generalized estimating equation linear regressions accounting for clustering of longitudinal observations within person, adjusted associations and 95% confidence intervals; Test type: Superiority; p = 0.11, Chi-squared; Slope = 0.35, 95% CI 2-sided [-0.07 to 0.78]

4. Secondary Outcome: Student Interviews to Qualitatively Assess Student Learning From All Educational Units and Changes in Student Perspectives, Behaviors, and Behavioral Intentions Related to Shellfish Harvesting.
Description: The investigators conducted interviews at the beginning and end of each semester's program (before and after all units). To analyze data, a codebook was generated using both inductive and deductive approaches. First, codes were identified based on major themes in the interview protocol and relevant to the TPB. Next, all transcripts were reviewed to identify further themes not captured in deductively developed codes. This grounded theory approach was important to identify new themes raised by participants. Data was coded and analyzed using Dedoose software. Here we report themes raised in post-program interviews. Participant quotations reflecting these themes can be found in the published paper from this study.
Time Frame: Post education (following the semester-long program) at 10 weeks.
Population: Differences between the participant numbers in the rows and the overall numbers are due to 30 total post-program interviews being conducted. Of the 50 participants in the study, 1 did not consent to participate in interviews. Of the 49 consented participants, interviews were conducted with 37 participants at the start of the program and 30 participants at the end of the program. Fewer interviews were conducted than the number of those consented because of scheduling and attendance constraints.
Measure: Count of Participants; unit: Participants
Arm/Group | Middle School Education Program
Number analyzed (Participants) | 30
Participants
  Some/ high knowledge of PSP | 26
  Some/ high knowledge of risk reduction strategies | 20
  Some/ high knowledge of SEATOR resources | 28

5. Secondary Outcome: Follow-up Student Assessment Questionnaire of Student Learning to Assess Lasting Behavioral Changes From Intervention Participation.
Description: The investigators will follow up with participants one year after participation in the educational program to assess whether participants have had any behavior changes related to subsistence shellfish consumption, measured using Likert scale questions. Likert-scale responses ranged from disagree (1) to agree (5).
Time Frame: Data collection one year following participation in the educational program.
Population: When we closed the study, only 7 participants had completed the program at least one year prior and were available for one year post-program recontact. Of these 7 participants, 4 completed the follow-up survey.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Middle School Education Program
Number analyzed (Participants) | 4
Scores on a scale
  7: I have participated in clam harvesting | 5 (0)
  8: Learning clam safety I am more willing to clam | 4.75 (0.5)
  15: I intend to check website to decide to clam | 5 (0)
  16: I have used website to inform decision to clam | 3.5 (1.9)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from participant study enrollment through study completion, which was approximately 10 weeks (or one educational semester) following enrollment.
Groups:
- Middle School Education Program: The education intervention centers around teaching children about local traditional ecological knowledge and traditional harvesting and gathering practices, including those for shellfish.
Arm/Group | Middle School Education Program
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/29/NCT05247229/Prot_SAP_ICF_000.pdf